CLINICAL TRIAL: NCT02508623
Title: Effect of Administration "Add on" of Rifaximin on Portal Hypertension of Patients With Liver Cirrhosis and Esophageal Varices in Standard Therapy With Propranolol
Brief Title: Effect of Administration of Rifaximin on the Portal Pressure of Patients With Liver Cirrhosis and Esophageal Varices
Acronym: ERASE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Piero Amodio, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3250/AO/14; 2014-000102-35 (EudraCT Number)
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: Portal hypertension; liver cirrhosis; Rifaximin
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental): Rifaximin 550 mg 1 tablet BID for 60 days
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Placebo 1 tablet BID for +60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 550 mg tablet BID for 60 days
  Arms: Rifaximin
Drug: Placebo — Placebo 1 tablet BID for 60 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether the add of Rifaximin in patients with liver cirrhosis and esophageal varices treated with a standard therapy with beta blockers, leads to a significant reduction of portal hypertension.

DETAILED DESCRIPTION:
It is well recognized that the gut flora may play an important role in the development of complications of liver cirrhosis, such as hepatic encephalopathy (HE), spontaneous bacterial peritonitis (SBP) and variceal bleeding, which are are directly caused or aggravated by the translocation of enteric bacteria or their products into the blood of cirrhotic patients.Preliminary studies have shown that selective intestinal decontamination appears to ameliorate the hyperdynamic circulatory state of cirrhosis. The investigators hypothesize that a modulation of gut microbiota by administering a non-adsorbable antibiotic, in addition to beta-blockers, can be a safe strategy to reduce the portal pressure, influencing favorably hemodynamics of portal circulation. Thus, the purpose of this study is to evaluate if in patients with liver cirrhosis and esophageal varices at high risk of bleeding, Rifaximin, administered in addition to standard therapy with beta - blockers (propranolol), for a time of 60 days: leads to a significant reduction of Hepatic Venous Pressure Gradient (it will be assessed by hepatic vein catheterization), 2) modify the intestinal flora in favor of specific families of bacteria (it will be assessed by fecal microbiota analysis), 3) change systemic inflammatory responses (it will be assessed by serum pro-inflammatory cytokines) 4) change in cognitive functions (it will be assessed by neuropsychological and electroencephalogram evaluations).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis (based on clinical, biochemical and radiological criteria with or without liver biopsy)
* Presence of esophageal varices at high risk of bleeding
* Hepatic Venous Pressure Gradient > 12 mmHg.
* 19≤ age ≤75
* Informed Consent

Exclusion Criteria:

* Patients already treated with beta blockers
* Treatment with systemic antibiotics and/or non-absorbable intestinal antibiotics in the previous two weeks
* Bacterial infection, spontaneous bacterial peritonitis
* overt hepatic encephalopathy in the last week
* active gastrointestinal bleeding, or in the last week
* active alcoholism or drug abuse in last 3 weeks
* Acute Alcoholic Hepatitis
* Hepatocellular carcinoma or other neoplasm
* significant coronary artery disease (angina NYHA III/IV), congestive heart failure (NYHA III/IV), relevant cardiomyopathy, history of myocardial infarct within the last 12 months
* Contraindications to the administration of beta blockers; allergy to Rifaximin
* Pregnancy or breastfeeding
* Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change of Hepatic Venous Pressure Gradient | Time 0 and after 60 days
  At Time 0 and after 60 days all patients will underwent hepatic vein catheterization to obtain the Hepatic Venous Pressure Gradient. Treatment response is defined as a decrease from baseline in the hepatic venous pressure gradient of at least 20% or less than 12 mmHg

SECONDARY OUTCOMES:
Modification of fecal bacteria | Time 0 and after 60 days
  Both at time 0 and after 60 days, samples of 3 mL of faeces produced within 6 hours will be collected and frozen at -80° for the analysis of the gut microbiota (the samples will be stored at -80°C). Gut microbiota will be studied through sequencing of hyper-variable regions of the 16S Ribosomal Ribonucleic Acid gene.
Change of systemic inflammatory response | Time 0 and after 60 days
  Both at time 0 and after 60 days, the storage of a serum sample at -80 ° for the assay of proinflammatory cytokines will be done.
Change of cognitive function | Time 0 and after 60 days
  Cognitive function will be assessed at time 0 and after 60 days by neuropsychological and neurophysiological measures. Neuropsychological investigation will be performed using the Italian version of the Psychometric Hepatic Encephalopathy Score that and with the Animal Naming Test (number of animals named in 60 sec). Neurophysiological investigation will be done by Emotiv Electroencephalogram equipment. Spontaneous closed-eyes rest activity will be recorded by a 14 channels plus 2 references offering optimal positioning for accurate spatial resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Amodio, Principal Investigator — University of Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Italy, Italy